CLINICAL TRIAL: NCT06092723
Title: Effects of Lactococcus Lactics Subsp. Lactics, LY-66, Lactobacillus Plantarum, PL-02, and Combination LY-66+PL-02 Improves the Endurance and Explosiveness Exercise Performance on Healthy Human.
Brief Title: Effects of Probiotics Improves the Endurance and Explosiveness Exercise Performance on Healthy Human.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glac Biotech Co., Ltd (Industry)
Responsible Party: Principal Investigator, Hsieh-Hsun Ho, R & D director, Glac Biotech Co., Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LSHIRB21-042-A2
Record Dates: First submitted 2023-09-28; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Exercise Performance
Keywords: Probiotics; Intestinal flora; Exercise Performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lactococcus lactis subsp. lactis, LY-66 (Experimental): Subjects take two packs once a day, and make a 250 ml water solution for drinking.
  Interventions: Dietary Supplement: Probiotic 1,Lactococcus lactis subsp. lactis, LY-66
- Lactobacillus plantarum, PL-02 (Experimental): Subjects take two packs once a day, and make a 250 ml water solution for drinking.
  Interventions: Dietary Supplement: Probiotic 2,Lactobacillus plantarum, PL-02
- Lactococcus lactis subsp. lactis, LY-66+Lactobacillus plantarum, PL-02 (Experimental): Subjects take two packs once a day, and make a 250 ml water solution for drinking.
  Interventions: Dietary Supplement: Probiotic 3,Lactococcus lactis subsp. lactis, LY-66+Lactobacillus plantarum, PL-02
- Placebo (Placebo Comparator): Subjects take two packs once a day, and make a 250 ml water solution for drinking.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Subjects take two packs once a day, and make a 250 ml water solution for drinking.
  Arms: Placebo
Dietary Supplement: Probiotic 1,Lactococcus lactis subsp. lactis, LY-66 — Subjects take two packs once a day, and make a 250 ml water solution for drinking.
  Arms: Lactococcus lactis subsp. lactis, LY-66
Dietary Supplement: Probiotic 2,Lactobacillus plantarum, PL-02 — Subjects take two packs once a day, and make a 250 ml water solution for drinking.
  Arms: Lactobacillus plantarum, PL-02
Dietary Supplement: Probiotic 3,Lactococcus lactis subsp. lactis, LY-66+Lactobacillus plantarum, PL-02 — Subjects take two packs once a day, and make a 250 ml water solution for drinking.
  Arms: Lactococcus lactis subsp. lactis, LY-66+Lactobacillus plantarum, PL-02

SUMMARY:
This study may discover that supplementing with probiotics LY-66, PL-02 can promote exercise endurance, explosive power and reduce muscle inflammation index in healthy people.

DETAILED DESCRIPTION:
With the rise of people's health awareness and exercise habit in recent years, and the demand for the use of sports health food supplements has also increased. Probiotics are generally recognized as safe and helpful in digestion in the gastrointestinal tract. Previous animal experiments have found that probiotics LY-66, PL-02 are more effective in promoting the grip and exhausting exercise in mice. The purpose of this study is to further explore the effects of probiotics LY-66, PL-02 on promoting exercise endurance and explosive power in healthy people. This study is to compare supplementary samples with placebo and adopt a double-blind study design. 88 healthy adult males and females (non-sports players) aged 20-40 will be recruited, 44males and 44 females, with an average number of male and female subjects in each group, and they will be randomly assigned to the (A) placebo group, (B) LY-66 probiotic group, (C) PL-02 probiotics group, (D) LY-66/PL-02 doublet probiotics group. Supplemented one time a day, take 15 billion CFU of probiotics each time for 42 consecutive days. During the period of taking probiotics, squats and TABATA training were set for the subjects 2 days a week. From day 0 to day 42 of supplementation, subjects in each group were tested physical fitness and cardiorespiratory endurance every 14 days. On the 21th days, the explosiveness of muscle strength in each group was tested with Wingate. On the 42nd day, the exercise endurance test, NGS and GC-MS technology was used to detect the fecal microbiota and SCFA(Short-chain fatty acids) in each group, body inflammation index of each group were tested and use questionnaire to evaluate subjective experience. This study may discover that supplementing with probiotics LY-66, PL-02 can promote exercise endurance, explosive power and reduce muscle inflammation index in healthy people.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult
2. Age 20-40
3. Not professional athletes

Exclusion Criteria:

1. The patient who Smoking.
2. The patient have cardiovascular disease
3. The patient have hyertension
4. The patient BMI>27
5. The patient have metabolic diseases
6. The patient have asthma
7. The patient who have experienced limb, neuromuscular, or exercise-related injuries within the past 6 months,.
8. The patient have taken anti-inflammatory or pain-relief medication in the past month,
9. The patient have consumed probiotic-related products will be excluded.
10. Students under the supervision of the principal investigator and individuals with conflicts of interest .

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Compare the enhancing endurance performance in sports. | before、Week6
  The Isometric Mid-Thigh Pull (IMTP) is a reliable and valid test that can be used to measure maximal force using a custom-made IMTP test device and a force plate. The measured parameters are Peak Force ( the maximum value of force)
Wingate Anaerobic test | before、Week 3、Week6
  Use an anaerobic power bicycle and sprint at full speed for 30 seconds. The measured parameters are Peak power (peak power output, which is the output during the test).
Compare muscle gain and fat loss. | before、Week 0、Week 2、Week4、Week6
  Use body fat meter to measure body composition.
Compare the enhancing explosive power performance in sports. | before、Week 3、Week6
  Using a force plate and an infrared high-speed camera, a light ball was installed on the subject, and the subject was asked to jump three times at their maximum ability. The maximum jumping force is calculated based on the distance of optical capture displacement.
Changes in maximal oxygen uptake(VO2 max) | before、Week6
  When the heart rate reaches 170 beats per minute, start collecting gas until exhaustion. The collected gas is used to calculate VO2max through a gas analyzer. The standard for judging exercise exhaustion is that two of the following three conditions are met:
  (A) The heart rate reaches the maximum heart rate (maximum heart rate = 220 - age).
  (B) The subject's respiratory exchange rate reaches 1.1. (C) The subject's self-motivated expression of exercise is above 18.

SECONDARY OUTCOMES:
Changes in sleep quality | Week0、Week3、Week6
  The ratio of deep sleep to light sleep in sleep was record before and during the trial. Changes in PITTSBURGH SLEEP QUALITY INDEX (PSQI) scores were record at before and after intervention. The minimum value is "0" and maximum value is "72", higher scores mean a worse outcome.
Changes in stool form. | Before、Week 6
  Record the stool form at before anf week 6.Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 indicating lack of dietary fiber, and 6 and 7 indicate diarrhoea.(Type 1: Separate hard lumps, like nuts (difficult to pass)、Type 2: Sausage-shaped, but lumpy、Type 3: Like a sausage but with cracks on its surface、Type 4: Like a sausage or snake, smooth and soft (average stool)、Type 5: Soft blobs with clear cut edges、Type 6: Fluffy pieces with ragged edges, a mushy stool (diarrhea)、Type 7: Watery, no solid pieces, entirely liquid (diarrhea))
Changes in immune Index (pg/ml). | before the exhaustive exercise and 3 hours、24hours、48hours after the exhaustive exercise.
  Exercise program to induce muscle fatigue and soreness This exercise program for inducing muscle fatigue and soreness involves 100 repeated jumps. Divide 100 jumps into 10 groups, 10 times each, and complete one jump in 4 seconds each time.
  Changes in Creatine kinase、Cortisol、IL-6 were assessed before the exhaustive exercise and 3 hours、24hours、48hours after the exhaustive exercise.
Changes in immune Index (pg/ml). | Before、Week 6
  Changes in AST、ALT、blood urea nitrogen, creatinine, uric acid, ketone bodies, total protein, total cholesterol, triglycerides, high-density lipoprotein, low-density lipoprotein, glucose, serotonin, melanin and short-chain fatty acid concentrations were assessed before and week 6.

CONTACTS AND LOCATIONS:
Locations (1):
- Glac Biotech Co., Ltd., Tainan, Taiwan